CLINICAL TRIAL: NCT06736652
Title: Operational Performance Effects and Neurophysiology in Partial Gravity
Acronym: OPEN-PG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gary E. Strangman, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022P003142
Record Dates: First submitted 2024-05-30; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-05

CONDITIONS: Physiological Stress
Keywords: partial gravity; microgravity; neurophyisology; behavioral performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main study arm (Experimental): All subjects perform the same activities (described in the protocol), but in different orders for counterbalancing purposes.
  Interventions: Other: Parabolic flight

INTERVENTIONS:
Other: Parabolic flight — Preflight each individual was exposed to the 3 Other Interventions and monitored for changes in behavioral performance and neurophysiological responses. In-flight the same monitoring was conducted during partial-gravity (0.25, 0.5. 0.75g) and microgravity (~0g).
  Other Names: Galvanic vestibular stimulation; Vection; Head tilts

SUMMARY:
Aim 1: Characterize and quantify changes in operationally-relevant sensorimotor and vestibular performance as a function of gravitational load.

Aim 2: Characterize and quantify changes in physiology-particularly in brain function and autonomic activation during behavioral performance-as a function of gravitational load.

Aim 3: Develop a model to predict behavioral performance and neurophysiological responses under different gravitational loads based on preflight ground testing data.

(Hyp1) The investigators predict a monotonic but non-linear relationship between operational performance (grappling / postural sway) and gravitational load, with larger departures from 1g leading to more impaired performance.

(Hyp2) The investigators predict a similar relationship between gravity load and physiological measures, with larger departures from 1g leading to larger changes in prefrontal and vestibular cortex, and autonomic nervous system activation.

(Hyp3) Ground-based challenges to the vestibular system will induce detectable postural sway and neurophysiological responses. The amplitude of these responses and/or adaptation rates to the challenges (i.e., indicators of individual "sensitivity" to such provocations) will (3a) help predict neurophysiological responses in-flight, and (3b) help predict behavioral performance in flight.

DETAILED DESCRIPTION:
Physiological Recording Setup: Dr. Strangman's NINscan devices support 64-channel near-infrared spectroscopy (NIRS), plus multiple electrophysiological and related measurements. The NIRS pad will be positioned to span the right lateral prefrontal cortex to parietal vestibular cortex, given the typical right-lateralization of the working memory, spatial processing, and vestibular brain functions under investigation 2, 7, 22. A multi-separation probe will help remove scalp and skull hemodynamic interference in the fNIRS signal 25, 27. Accelerometers will be placed on the head and sacrum to detect motion artifacts and sway. Planned additional sensors will include EEG over prefrontal and parietal locations (e.g., International Standard locations Fz/F7/P3 14) plus two electrooculography sensors to measure eye movements, 1 ECG sensor for cardiac activity, two facial electromyography sensors, skin temperature, and electrodermal activity (EDA). Skin markers may be used to facilitate flight-day setup.

Phase 0: On-Ground (Preflight) Subject Training Preflight Training: Preflight training will focus on the following: (i) self-deployment of the NINscan system, and performance of (ii) the ROBoT-r task, and (iii) postural sway. On Day 1, subjects will participate in a ~90-min Familiarization session, followed by a 1st ~90-min Training session. On Day 2, subjects will perform the 2nd Training session. Each Training session will include a 10-min resting-state baseline period during which subjects will sit quietly with their eyes-open (to practice and to provide baseline data on e.g. functional connectivity, intracranial pulsatility, BP, EEG, and EDA), followed by performance of ROBoT-r and postural sway tasks.

NINscan: Familiarization will include instruction on the hardware, self-deployment, safe operation, and basic troubleshooting. For training sessions, participants will self-deploy the device, including attachment of all brain and physiologic sensors, and collect data while performing ROBoT-r and postural sway tasks, with instructor supervision throughout.

ROBoT Docking: Participants will perform ROBoT-r training via our published approach 5, including instruction on (i) system components, (ii) performance criteria, and (iii) basic troubleshooting. During training sessions, participants will deploy ROBoT-r and perform a full session (12 runs) while standing on a posturography platform and wearing NINscan.

Postural Sway: During familiarization, participants will learn to safely maintain upright stance on a Zibrio-Pro (Zibrio, Houston, TX) computerized posturography platform. This will involve standing upright with head erect, arms next to their body, with their feet on the platform at shoulder width. The subjects will then be familiarized with the vestibular challenges: (1) performance of ±20⁰ dynamic head pitch-tilt oscillations at 0.33 Hz paced by an audible tone 12, 13, (2) viewing the circularly-rotating visual stimulus and reporting vection sensations, and (3) the Galvanic vestibular stimulation system. The Training sessions will not involve any vestibular challenges, just practice with the balance/posturography testing.

Phase 1: On-Ground (Preflight) Baseline Data Collection Ground Baseline Data Collection (BDC): After training, participants will participate in three baseline data collection procedures, spread over 3 days to minimize interference effects. Each session will include a rest recording, postural sway, docking, and one of our three neurovestibular challenges (counterbalanced to minimize potential order effects).

BDC Rest Recording: Each participant will fill out the Motion Sickness Susceptibility Questionnaire (MSSQ) first 3. They will then self-deploy the NINscan recording device (with experimenter oversight) to wear throughout the BDC period, starting with a 10-min rest recording.

BDC Postural Sway: Participants will then perform the postural sway task (above), using NINscan while standing on the computerized posturography platform to obtain baseline sway at 1g.

BDC Docking: Next, participants will perform a set of 12 ROBoT-r runs. Brief rest periods will occur between runs. This will provide baseline data on operationally relevant task performance in 1g.

BDC Neurovestibular Challenges: For our predictive models (Aim 3), the investigators will assess participants' preflight responses to three neurovestibular challenges, each based on a distinct type of sensory input. NINscan recordings will record throughout each exposure period. Challenges will be provided on each of 3 consecutive days, in counterbalanced orders. A Likert-style motion sickness scale (0-10) will be used to assess acute symptoms 11, while the Motion Sickness Symptoms Questionnaire (MSSQ) will be administered before and after each data collection session. All vestibular challenges will be performed while standing on the Zibrio posturography plate. Postural Sway recordings will start 2 min prior to vestibular challenges, and continue until 2 min after completion of challenges, each as described below.

1. Galvanic vestibular stimulation (GVS) and adaptation (electrical input) 1, 8, 9. Participants standing on the posturography platform will undergo 25s periods of GVS over the mastoid processes (interleaved with rest periods) using a pseudorandom current waveform stimulus consisting of a sum-of-sines (0.16, 0.33, 0.43, 0.61 Hz) with a peak amplitude of 5 mA. These parameters are designed to replicate the postflight sensorimotor experience of astronauts 1. Three cycles of twelve alternations will be presented every 15 minutes for a total of 45 minutes to assess adaptation.
2. Roll-vection and adaptation (visual input, non-otolith) 10, 15, 23. Standing subjects will view a central fixation cross on a computer monitor. A sparse field of stars will be rotated around the central point (60 deg/s), while the stars themselves rotate in the same direction to enhance the vection effect (60 deg/s) 10. Participants press a key whenever vection (self-rotation in the opposite direction of the visual stimulus) is perceived, and release it when the perception ceases 10. Stimulus periods will be 25s long, interleaved with 25s periods of a blank screen. During the blank screens, participants will verbally report the strength of the vection perception on a 0-100 scale (0=none, 50=the same vection as perceived in an initial, pretest single exposure to a globally-rotating stimulus 10). Again, three cycles of twelve stimulus/blank exposures will be presented every 15 minutes for a total of 45 minutes to assess adaptation.
3. Oscillatory head pitch (mechanical input) 12, 13. Standing participants will either hold their head erect and static (HS), or perform continuous ±20 dynamic pitch oscillations (head dynamic, HD) at 0.33 Hz paced by an audible tone transmitted through lightweight headphones. White noise supplied through headphones will mask external auditory orientation cues. Three cycles of 12 HS and HD alternations will be performed during 45 minutes to assess adaptation.

Phase 2: Flight Data Collection

Flight testing: On flight day, participants will be pre-instrumented on the ground for rapid NINscan deployment. Anti-motion sickness medication will not be allowed for these participants, as it interferes with the neurovestibular measurements the investigators are making. Participants board the Airbus A310 ZERO-G and fasten seatbelts for takeoff. After takeoff, the pilots fly the aircraft to a specific air zone where the parabolas will take place. With other members of the participant's group and the instructor, participants will then move to the area of the cabin. Participants will receive instructions from Novespace to maintain safety during the parabolic flight. Upon reaching level flight, participants will don NINscan, start NINscan recording, and initialize the ROBoT-r equipment. Each participant will stand on a computerized posturography platform and perform two tasks during the 10 parabolas at each gravitational load (and for equivalent time periods during level flight at 1g): (1) operationally-relevant ROBoT-r task for the first 7 parabolas, and (2) postural sway assessment on the last 3 parabolas. As currently scheduled, there will be two flights for each participant. The first flight will include all n=12 participants and fly 31 parabolas, the first of which is for general orientation. Groups of 4 subjects will simultaneously perform the described tasks for 10 parabolas, and then they will switch places with the next group of 4 subjects. On the second flight for each participant, the plane will fly 31 parabolas again, the first being for orientation. After that, 3 sets of 10 parabolas will be flown, each set at a different gravity level (nominally 0.25, 0.5 and 0.75g). Participants will perform tasks during all three groups of 10 parabolas, identical to the 10 parabolas at 0. An additional period of level flight will be performed where participants again perform the same tasks on the same timeline, but at 1g. Participants will be closely monitored throughout by a dedicated experimenter and/or harnessed (as required by Novespace) to ensure safety.

If a participants agrees to the photo/video clause in the informed consent, photos/videos of their participation may be conducted during the flight. These will either be taken from behind the participant, or any facial features will be blurred and prior to use in any presentation or publication form.

There will be no post-flight activities for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 30-55-year-olds
* Willingness and ability to participate in flights without motion sickness medications.
* Any Novespace requirements

Exclusion Criteria:

* Failure to meet medical criteria and provide certification of fitness for flight to NOVESPACE (i.e., NOVESPACE Parabolic Flight Medical Aptitude Certificate) completed by their medical doctor or an Authorized Medical Examiner
* Certain heart and lung conditions
* Dizziness
* Certain inner ear conditions
* Severe motor disability or impaired bone density
* Psychosis
* Mental disability prohibiting emergency evacuation.
* Epilepsy
* Certain neurological diseases
* Fear of heights/flying
* Debilitating anxiety and panic attacks
* Claustrophobia
* Women who are pregnant
* Certain gastrointestinal conditions
* Those taking certain medications. An individual's overall medical fitness for flight is assessed and certified by a medical doctor or Authorized Medical Examiner.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
ROBoT-r | 10 days
  Operationally-relevant track-and capture behavioral measures
Postural stability | 10 days
  Operationally-relevant standing balance measure

CONTACTS AND LOCATIONS:
Locations (1):
- NoveSpace, Mérignac, France

IPD SHARING:
Plan to Share IPD: Yes
All IPD from this project will be anonymized IPD and shared. Data will be coded with a key only available to the Principal Investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available by the end-date of the funded project (estimated 5/31/2026) and be retained indefinitely.
Access Criteria: Researchers will be allowed to request the data from the NLSP through their website: https://nlsp.nasa.gov/explore/page/home. NASA will be responsible for vetting requests and providing the data as requested.
URL: https://nlsp.nasa.gov/explore/page/home